CLINICAL TRIAL: NCT05815797
Title: The Safety and Effects of Using Shuiniujiao Dihuang Decoction With Variation for the Treatment of Psoriasis: A Double-blind, Randomized, Placebo-Controlled Trial
Brief Title: Shuiniujiao Dihuang Decoction With Variation for the Treatment of Psoriasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMDF Psoriasis Study
Record Dates: First submitted 2023-02-21; First posted 2023-04-18 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDD Formula (Experimental): Subjects will receive SDD Formula granules (37g twice daily) for 12 weeks.
  Interventions: Drug: SDD formula
- Placebo (Placebo Comparator): Subjects will receive placebo granules (37g twice daily) for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SDD formula — SDD formula consists of 23 herbal medicines
  Arms: SDD Formula
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Psoriasis is an inflammatory skin disease with huge negative impact on the quality of life of the patients, and has an overall prevalence of 2% to 3% in the general population. Plaques psoriasis is the most common type of the disease and presents red, well demarcated, and silvery plaques mainly localized in the umbilical and lumbosacral area as well as in the elbows, knees, and scalp.

Currently, pharmacological treatments such as retinoids, corticosteroids, vitamin D analogs and biologics remain the main options for most psoriasis patients. However, side effect and high cost barred many ordinary psoriasis patients from benefiting from the treatments.

A Chinese medicine formula "Shuiniujiao Dihuang Decoction with Variation (SDD)" was prescribed by Prof. Lin for many years and observed to be effective in relieving psoriasis patients' clinical manifestations.

In this study, subjects with psoriasis will be randomized into treatment group of "SDD" or placebo group for 12 weeks.

DETAILED DESCRIPTION:
Psoriasis is an inflammatory skin disease with huge negative impact on the quality of life of the patients, and has an overall prevalence of 2% to 3% in the general population. Plaques psoriasis is the most common type of the disease and presents red, well demarcated, and silvery plaques mainly localized in the umbilical and lumbosacral area as well as in the elbows, knees, and scalp. The major histological features of psoriasis include epidermal hyperplasia with aberrant keratinocyte differentiation, pronounced inflammatory cell infiltration and increased vascularization. Currently, pharmacological treatments such as retinoids, corticosteroids, and vitamin D analogs remain the main options for most psoriasis patients. However, the efficacy of conventional drugs is limited because of adverse side effects and the development of pharmacoresistance. Recently, biologics have become available for the treatment of acute and subacute plaque psoriasis with excellent response rate. However, the high costs involved with the biologics have barred many ordinary psoriasis patients from benefiting from this new class of anti-psoriatic medication.

Natural products are valuable sources in novel drug development. Shuiniujiao Dihuang Decoction with Variation (SDD) is an empirical formula of the Principal Investigator (Prof. Zhi-Xiu Lin), a highly experienced Registered Chinese Medicine Practitioner and Chinese medicine dermatologist working at the School of Chinese Medicine, The Chinese University of Hong Kong. SDD has been prescribed in clinic in Hong Kong for many years and observed to be effective in relieving psoriasis patients' clinical manifestations. SDD contains 23 Chinese herbal medicines, including Rehmanniae Radix (Dihuang), Bubali Cornu (Shuiniujiao), Paeoniae Radix Rubra (Chishao), Moutan Cortex (Mudanpi), Scrophulariae Radix (Xuanshen), Ophiopogonis Radix (Maidong), etc. The formula is composed of herbal medicines that can eliminate pathogenic heat, expel blood stasis and dampness, nourish yin, and have antipruritic effect.

A randomized, double-blinded, placebo-controlled trial will be conducted to evaluate the efficacy of SSD on psoriasis patients. Clinical evidence for the anti-psoriatic effects of SSD is a necessary step towards developing this Chinese medicine formula into an anti-psoriatic pharmaceutical agent.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate chronic plaque psoriasis (PASI score 3 to 12).
* Willingness to give informed consent.

Exclusion Criteria:

* Pustular or generalized erythrodermic psoriasis.
* Psoriatic arthritis with syndrome of spleen-kidney yang deficiency according to Chinese medicine theory.
* Systemic therapy for psoriasis 6 months prior to baseline.
* Use topical medications for psoriasis 14 days prior to baseline such as retinoids, corticosteroids, vitamin D analogues, tazarotene and tacrolimus.
* Has taken any antibiotics, probiotics and prebiotics 30 days prior to baseline.
* UV light therapy 30 days prior to baseline.
* Clinically significant laboratory abnormality in blood, liver or renal functions (≥1.5 times the upper limit of reference range).
* History of allergy to Chinese herbs.
* Known pregnant or lactation, or have a plan to conceive in 6 months.
* Known active gastric or duodenal ulcer, or severe arrhythmia.
* Unwillingness to comply with study protocol.
* Any other condition that in the opinion of the investigators could disadvantage the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) | Week 12
  The change in Psoriasis Area and Severity Index (PASI) score will be assessed. PASI scores include area involved, erythema, induration and scaling. It will be scored on a scale of 0 to 4 (0, meaning none; 1, mild; 2, moderate; 3, severe; and 4, very severe). It will be performed by 2 blinded assessors who have been trained. Four main areas were assessed for calculation of the PASI scores: the head, the trunk, the upper extremities, and the lower extremities, corresponding to 10%,20%,30%, and 40% of the total body area, respectively. The maximum score for PASI is 72.
Static Physician Global Assessment score (sPGA) | Week 12
  Participants are requested to expose their skin thoroughly before the photographs are taken at each visit. The sPGA is an investigator-rated assessment of overall disease severity to be evaluated on a 5-point scale, where 0=clear and 4=severe. The severity of erythema, scaling, and plaque are considered for assessment. It will be performed by 2 blinded assessors who have received training.

SECONDARY OUTCOMES:
Constitution in Chinese Medicine Questionnaire (Hong Kong Version) | Week 12
  The 60-item Constitution in Chinese Medicine Questionnaire (CCMQ) Hong Kong version will be used to assess the body constitution (BC) in Chinese medicine of subjects. According to Chinese medicine theory, there are 9-type of BC: gentleness (8 Items), Qi-deficiency (8 Items), Yang-deficiency (7 Items), Yin-deficiency (8 Items), phlegm-wetness (8 Items), wetness-heat (6 Items), blood-stasis (7 Items), Qi-depression (7 Items), and special diathesis (7 Items). Subjects will have to score on a 5-point Likert scale for each item where 1=never and 5=for most of the time. A final score for each BC will be calculated according to the scoring algorithm. A higher score in the CCMQ BC scale indicates a higher likelihood of the specific BC type, and a score of 30 is set as threshold for case definition. Coexistence of multiple imbalanced BC types is possible which is consistent with the Chinese medicine theories.
Chinese Medicine symptom pattern | Week 6
  A structural designed record form will be completed by Chinese medicine practitioner (CMP) to record the signs and symptoms of the subjects, which includes but not limited to spirit, skin condition, joints condition, sleep condition, tongue and pulse condition. A final symptom pattern will be decided by the CMP according to the form by Chinese medicine theory.
Chinese Medicine symptom pattern | Week 12
  A structural designed record form will be completed by Chinese medicine practitioner (CMP) to record the signs and symptoms of the subjects, which includes but not limited to spirit, skin condition, joints condition, sleep condition, tongue and pulse condition. A final symptom pattern will be decided by the CMP according to the form by Chinese medicine theory.
Chinese Medicine symptom pattern | Week 18
  A structural designed record form will be completed by Chinese medicine practitioner (CMP) to record the signs and symptoms of the subjects, which includes but not limited to spirit, skin condition, joints condition, sleep condition, tongue and pulse condition. A final symptom pattern will be decided by the CMP according to the form by Chinese medicine theory.
Psoriasis Area and Severity Index (PASI) | Week 6
  The change in Psoriasis Area and Severity Index (PASI) score will be assessed. PASI scores include area involved, erythema, induration and scaling. It will be scored on a scale of 0 to 4 (0, meaning none; 1, mild; 2, moderate; 3, severe; and 4, very severe). It will be performed by 2 blinded assessors who have been trained. Four main areas were assessed for calculation of the PASI scores: the head, the trunk, the upper extremities, and the lower extremities, corresponding to 10%,20%,30%, and 40% of the total body area, respectively. The maximum score for PASI is 72.
Psoriasis Area and Severity Index (PASI) | Week 18
  The change in Psoriasis Area and Severity Index (PASI) score will be assessed. PASI scores include area involved, erythema, induration and scaling. It will be scored on a scale of 0 to 4 (0, meaning none; 1, mild; 2, moderate; 3, severe; and 4, very severe). It will be performed by 2 blinded assessors who have been trained. Four main areas were assessed for calculation of the PASI scores: the head, the trunk, the upper extremities, and the lower extremities, corresponding to 10%,20%,30%, and 40% of the total body area, respectively. The maximum score for PASI is 72.
Static Physician Global Assessment score (sPGA) | Week 6
  Participants are requested to expose their skin thoroughly before the photographs are taken at each visit. The sPGA is an investigator-rated assessment of overall disease severity to be evaluated on a 5-point scale, where 0=clear and 4=severe. The severity of erythema, scaling, and plaque are considered for assessment. It will be performed by 2 blinded assessors who have received training.
Static Physician Global Assessment score (sPGA) | Week 18
  Participants are requested to expose their skin thoroughly before the photographs are taken at each visit. The sPGA is an investigator-rated assessment of overall disease severity to be evaluated on a 5-point scale, where 0=clear and 4=severe. The severity of erythema, scaling, and plaque are considered for assessment. It will be performed by 2 blinded assessors who have received training.
Psoriasis-involved body surface area (BSA) | Week 6
  BSA represents the affected skin surface. It is an objective measure of psoriasis severity. The head, the upper extremities, the trunk, and the lower extremities, corresponding to 10%,20%,30%, and 40% of the total body area, respectively. The range of BSA is 0-100. It will be performed by 2 blinded assessors who have received training by Dr Steven Loo.
Psoriasis-involved body surface area (BSA) | Week 12
  BSA represents the affected skin surface. It is an objective measure of psoriasis severity. The head, the upper extremities, the trunk, and the lower extremities, corresponding to 10%,20%,30%, and 40% of the total body area, respectively. The range of BSA is 0-100. It will be performed by 2 blinded assessors who have received training by Dr Steven Loo.
Psoriasis-involved body surface area (BSA) | Week 18
  BSA represents the affected skin surface. It is an objective measure of psoriasis severity. The head, the upper extremities, the trunk, and the lower extremities, corresponding to 10%,20%,30%, and 40% of the total body area, respectively. The range of BSA is 0-100. It will be performed by 2 blinded assessors who have received training by Dr Steven Loo.
Impact of Psoriasis Questionnaire (IPSO) | Week 12
  The change in Impact of Psoriasis Questionnaire (IPSO) score will be assessed. IPSO is a validated 16-item psoriasis-specific instrument for quality of life of psoriasis patients. The IPSO is intended predominantly to assess the psychosocial impact of psoriasis on patient's lives. The IPSO uses an ordinal rating scale, with responses of 'none', 'some', 'moderately', 'quite a bit' and 'extremely' scored 1, 2, 3, 4 and 5, respectively. The scores for item 4 were reversed. The higher the summed score, the greater the impact experienced due to psoriasis.
Short Form 36 survey (SF36) | Week 12
  The change in the score of quality of life using Short Form 36 survey (SF36) will be assessed. SF36 is generic instrument to measure general health status that is complementary to those derived from dermatological questionnaires. It will be used to assess the patient's health status using 8 different dimensions including vitality, physical functioning, bodily pain, general health perceptions, role limitations due to physical health, role limitations due to emotional health, social role functioning and mental health. The possible score ranges from 0 to 100 points whereby 0 points represent the greatest possible limitation of health, while 100 points represent the absence of health restrictions.
Psoriasis Itch Visual Analog Scale (Itch VAS) | Week 12
  Psoriasis itch VAS is a validated tool to assess treatment benefit of plaque psoriasis. It was developed to measure itch intensity within the last 24 hours. A horizontal line with a length of 100mm is to be used to represented the range of itch intensity from 0 (no itch at all) to 100 (worst itch you can imagine). Subjects rated the maximal intensity of itch during the previous 24 hours by putting a vertical mark through the horizontal line at the the spot he/she felt best reflected their maximal itch intensity.
Use of rescue therapy | Day 0 to Week 18
  The frequent use of rescue therapy during study period
Adverse events | Day 0 to Week 18
  Adverse events related to study treatment
Serum markers (IL-17, IL-22) | Week 6
  The changes in levels of serum markers IL-17, IL-22
Serum markers (CRP ) | Week 6
  The changes in levels of serum markers C-reactive protein (CRP)
Serum markes (BD2) | Week 6
  The changes in levels of serum marker Beta-Defensin 2 (BD2).
Serum markers (IL-17, IL-22) | Week 12
  The changes in levels of serum markers IL-17, IL-22
Serum markers (CRP) | Week 12
  The changes in levels of serum markers C-reactive protein (CRP)
Serum markers (BD2) | Week 12
  The changes in levels of serum marker Beta-Defensin 2 (BD2).
Oral and Gut microbiota composition in saliva and stools | Week 12
  Saliva and stool specimen will be collected at baseline and week 12 (+/-4 days) for gut microbiota assessments.
Gene expression of serum inflammatory factors | Week 6
  The changes in gene expression of serum inflammatory factors will be assessed by using the blood sample taken on baseline, week 6 and week 12. Analysis of such item could help to explore the effect mechanism of investigating medicinal product on gene expression of serum inflammatory factors on psoriasis patients.
Gene expression of serum inflammatory factors | Week 12
  The changes in gene expression of serum inflammatory factors will be assessed by using the blood sample taken on baseline, week 6 and week 12. Analysis of such item could help to explore the effect mechanism of investigating medicinal product on gene expression of serum inflammatory factors on psoriasis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu LIN, PhD, Principal Investigator — Hong Kong Institute of Integrative Medicine